CLINICAL TRIAL: NCT01098747
Title: Evaluation Of The Efficacy Of A Novel Ibuprofen Formulation In The Treatment Of Post-Surgical Dental Pain: Study I
Brief Title: Study Evaluating A Novel Ibuprofen Formulation In The Treatment Of Dental Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AH-09-10
Record Dates: First submitted 2010-04-01; First posted 2010-04-05 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-07

CONDITIONS: Pain
Keywords: Pain following third molar extraction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental)
  Interventions: Drug: Novel Ibuprofen
- Treatment B (Active Comparator)
  Interventions: Drug: Standard Ibuprofen
- Treatment C (Active Comparator)
  Interventions: Drug: Standard Ibuprofen
- Treatment D (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Novel Ibuprofen — Single-dose of novel ibuprofen (equal to 400 mg ibuprofen)
  Arms: Treatment A
Drug: Standard Ibuprofen — Single-dose of standard ibuprofen (400mg)
  Arms: Treatment B
Drug: Standard Ibuprofen — Single-dose of standard ibuprofen (400mg)
  Arms: Treatment C
Drug: Placebo — Single-dose of placebo
  Arms: Treatment D

SUMMARY:
This study will compare the pain relieving effect of a single-dose of a novel ibuprofen formulation to placebo and two formulations of standard ibuprofen in the treatment of post-surgical dental pain following "wisdom" tooth (third molar) removal.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy males and females 16 to 40 years of age
* Outpatients who have moderate to severe post-operative pain (confirmed by a Visual Analog Scale-Pain Severity Rating [VAS-PSR] score of at least 50 mm on a 100 mm VAS-PSR) following surgical extraction of two or more third molars, at least one of which must be a partial or complete bony mandibular impaction
* Use of only the following pre-operative medication(s)/anesthetic(s): topical benzocaine, a short acting parenteral (local) anesthetic (mepivacaine or lidocaine) with or without vasoconstrictor and/or nitrous oxide

Exclusion Criteria:

* Pregnancy or breast-feeding
* Alcohol or substance abuse
* Any serious medical or psychiatric disorder
* History of stomach ulcers, stomach bleed, or other bleeding disorders
* Use of a prescription or over-the-counter drug with which administration of ibuprofen or any other non-steroidal anti-inflammatory drug, acetaminophen, or hydrocodone is contraindicated (including: opioids, antipsychotics, antianxiety agents, or other central nervous system depressants[including alcohol])

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 335 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Jayawardena S, Leyva R, Kellstein D. Safety of a novel formulation of ibuprofen sodium compared with standard ibuprofen and placebo. Postgrad Med. 2015 Jan;127(1):33-7. doi: 10.1080/00325481.2015.993268. Epub 2014 Dec 15. PMID 25526232
- [Derived] Brain P, Leyva R, Doyle G, Kellstein D. Onset of analgesia and efficacy of ibuprofen sodium in postsurgical dental pain: a randomized, placebo-controlled study versus standard ibuprofen. Clin J Pain. 2015 May;31(5):444-50. doi: 10.1097/AJP.0000000000000142. PMID 25119511
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=AH-09-10&StudyName=Study%20Evaluating%20A%20Novel%20Ibuprofen%20Formulation%20In%20The%20Treatment%20Of%20Dental%20Pain

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Single oral dose of 2 placebo tablets.
- Ibuprofen Sodium: Single oral dose of 2 ibuprofen sodium 256 milligram (mg) tablets, equivalent to 400 mg ibuprofen.
- Ibuprofen (Advil): Single oral dose of 2 ibuprofen (Advil) 200 mg tablets (total dose of 400 mg ibuprofen).
- Ibuprofen (Motrin IB): Single oral dose of 2 ibuprofen [Motrin ibuprofen (IB)] 200 mg tablets (total dose of 400 mg ibuprofen).
Period: Overall Study
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil) | Ibuprofen (Motrin IB)
Started | 48 | 95 | 86 | 87
Completed | 48 | 95 | 86 | 87
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil) | Ibuprofen (Motrin IB) | Total
Number analyzed (Participants) | 48 | 95 | 86 | 87 | 316
Age Continuous [Mean (Standard Deviation); unit: Years] | 18.1 (1.6) | 18.6 (2.1) | 18.6 (2.3) | 18.4 (2.0) | 18.5 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 48 | 44 | 44 | 161
  Male | 23 | 47 | 42 | 43 | 155
Number of Participants with Pain Severity Score [Number; unit: Participants] — Pain severity score was assessed on a 4-point categorical scale. Total possible pain severity score range was 0 to 3, where 0 = none, 1 = mild, 2 = moderate and 3 = severe.
  Participants
    Moderate | 27 | 51 | 43 | 43 | 164
    Severe | 21 | 44 | 43 | 44 | 152

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of Pain Relief Rating and Pain Intensity Difference From 0-8 Hours (SPRID 0-8)
Description: SPRID: time-weighted sum of pain relief rating combined with pain intensity difference (PRID) over 8 hours. SPRID 0-8 score range: -8 (worst) to 56 (best). PRID: sum of Pain intensity differences (PID) and pain relief rating (PRR) at each time point. PRID score range: -1=worst to 7=best. PID: baseline pain severity score minus pain severity score at a given time point (pain severity score range 0=none to 3=severe; baseline score range 2=moderate to 3=severe). PID score range: -1(worst) to 3 (best). PRR: assessed on 5-point pain relief rating scale (0=No relief to 4=Complete relief).
Time Frame: 0 to 8 hours
Population: Intent-to-treat (ITT) population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium
Number analyzed (Participants) | 48 | 95
Units on a scale | 5.4 (14.1) | 29.8 (14.2)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; Treatment difference (Ibuprofen sodium - placebo) and 95 percent (%) confidence interval (CI):based on LS means from analysis of variance(ANOVA). Type I error controlled at 5% significance level (2-sided) by testing primary endpoints sequentially: Ibuprofen sodium (IBU Na) versus(vs.) Placebo for SPRID 0-8 then time to meaningful relief(TMR), IBU Na vs. IBU (Advil and Motrin IB) for TMR. If comparison at preceding step was significant only then subsequent comparisons were significant; Test type: Superiority or Other; p < 0.001, ANOVA — p-value was calculated using ANOVA model with treatment, baseline Pain Severity Rating (PSR) and gender terms; Least-square (LS) mean difference = 24.21, 95% CI 2-sided [19.32 to 29.09]

2. Primary Outcome: Time to Onset of Meaningful Relief
Description: Participants evaluated the time to meaningful relief by stopping a second stopwatch labeled 'meaningful relief' at the moment they first began to experience meaningful relief. Stopwatch was active up to 8 hours after dosing or until stopped by the participant, or rescue medication was administered.
Time Frame: 0 to 8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: Minutes
Groups:
- Ibuprofen (Advil + Motrin IB): Single oral dose of 2 ibuprofen (Advil) 200 mg tablets or Single oral dose of 2 ibuprofen (Motrin IB) 200 mg tablets.
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Minutes | NA [NA to NA] — Data was not summarized as median time to meaningful relief was greater than (>) 480 minutes (>8 hours) for placebo group and therefore 95% CI was not estimable. | 42.4 [38.5 to 46.6] | 55.3 [49.6 to 64.3]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; Hazard Ratio (HR) and corresponding 95% CI were calculated based on the Wald statistic from the proportional hazards (PH) model. Type I error controlled at 5% significance level (2-sided) by testing primary endpoints sequentially: IBU Na vs. Placebo for SPRID 0-8 then TMR, IBU Na vs. IBU (Advil and Motrin IB) for TMR. If comparison at preceding step was significant only then subsequent comparisons were significant; Test type: Superiority or Other; p < 0.001, Proportional hazards model — p-value was calculated using the PH model with treatment, baseline PSR and gender terms; Hazard Ratio (HR) = 12.80, 95% CI 2-sided [6.78 to 24.15]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model. Type I error controlled at 5% significance level (2-sided) by testing primary endpoints sequentially: IBU Na vs. Placebo for SPRID 0-8 then TMR, IBU Na vs. IBU (Advil and Motrin IB) for TMR. If comparison at preceding step was significant only then subsequent comparisons were significant; Test type: Superiority or Other; p < 0.001, Proportional hazards model — p-value was calculated using the PH model with treatment, baseline PSR and gender terms; Hazard Ratio (HR) = 1.59, 95% CI 2-sided [1.22 to 2.06]

3. Secondary Outcome: Time to Confirmed First Perceptible Relief
Description: Participants evaluated the time to first perceptible relief by stopping a stopwatch labeled 'first perceptible relief' at the moment they first began to experience any relief. Stopwatch was active up to 8 hours after dosing or until stopped by the participant, or rescue medication was administered. The first perceptible relief was considered confirmed if the participant also stopped the second stopwatch indicating meaningful relief.
Time Frame: 0 to 8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Minutes | NA [NA to NA] — Data was not summarized as median time to confirmed first perceptible relief was >480 minutes (>8 hours) for placebo group and therefore 95% CI was not estimable. | 16.4 [15.6 to 19.3] | 25.7 [22.2 to 29.1]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p < 0.001, Proportional hazards model — p-value was calculated using the PH model with treatment, baseline PSR and gender terms. Statistical testing was done at 5% significance level (2-sided); Hazard Ratio (HR) = 12.36, 95% CI 2-sided [6.51 to 23.46]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p < 0.001, Proportional hazards model — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.80, 95% CI 2-sided [1.38 to 2.34]

4. Secondary Outcome: Pain Relief Rating (PRR)
Description: PRR was evaluated at different time points during the study up to 8 hours after taking the study medication, and immediately before rescue medication was taken (if necessary). PRR was assessed on a 5-point categorical pain relief rating scale where 0=No relief to 4=Complete relief.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Units on a scale
  0.25 hours | 0.4 (0.6) | 0.7 (0.8) | 0.5 (0.7)
  0.5 hours | 0.5 (0.7) | 2.0 (1.1) | 1.5 (1.1)
  1 hour | 0.6 (1.0) | 2.9 (1.0) | 2.5 (1.1)
  1.5 hours | 0.7 (1.1) | 3.1 (1.0) | 2.8 (1.2)
  2 hours | 0.7 (1.2) | 3.1 (1.1) | 3.0 (1.2)
  3 hours | 0.7 (1.2) | 2.9 (1.2) | 3.0 (1.2)
  4 hours | 0.8 (1.3) | 2.8 (1.2) | 3.0 (1.2)
  5 hours | 0.7 (1.3) | 2.6 (1.3) | 2.8 (1.3)
  6 hours | 0.7 (1.2) | 2.3 (1.4) | 2.6 (1.4)
  7 hours | 0.5 (1.1) | 1.9 (1.4) | 2.3 (1.5)
  8 hours | 0.5 (1.1) | 1.7 (1.4) | 2.2 (1.5)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; 0.25 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.007, ANOVA — p-value was calculated using ANOVA model with treatment, baseline PSR and gender terms. Statistical testing was done at 5% significance level (2-sided); LS mean difference = 0.35, 95% CI 2-sided [0.10 to 0.60]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 0.25 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.010, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.24, 95% CI 2-sided [0.06 to 0.42]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Sodium; 0.5 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95 % CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.47, 95% CI 2-sided [1.10 to 1.84]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 0.5 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.53, 95% CI 2-sided [0.27 to 0.80]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen Sodium; 1 hour: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.22, 95% CI 2-sided [1.84 to 2.60]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 1 hour: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.006, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.39, 95% CI 2-sided [0.12 to 0.66]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; 1.5 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.39, 95% CI 2-sided [2.00 to 2.77]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 1.5 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.022, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.33, 95% CI 2-sided [0.05 to 0.60]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen Sodium; 2 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.39, 95% CI 2-sided [2.00 to 2.79]
Statistical Analysis 10: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 2 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.369, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.13, 95% CI 2-sided [-0.15 to 0.41]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen Sodium; 3 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.19, 95% CI 2-sided [1.78 to 2.60]
Statistical Analysis 12: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 3 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.420, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.12, 95% CI 2-sided [-0.42 to 0.17]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; 4 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.02, 95% CI 2-sided [1.58 to 2.45]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 4 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.151, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.23, 95% CI 2-sided [-0.54 to 0.08]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen Sodium; 5 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.88, 95% CI 2-sided [1.43 to 2.33]
Statistical Analysis 16: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 5 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.160, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.23, 95% CI 2-sided [-0.56 to 0.09]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen Sodium; 6 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.63, 95% CI 2-sided [1.16 to 2.10]
Statistical Analysis 18: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 6 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.055, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.33, 95% CI 2-sided [-0.67 to 0.01]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen Sodium; 7 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — p-value was calculated using ANOVA model with treatment, baseline PSR and gender PSR terms. Statistical testing was done at 5% significance level (2-sided); LS mean difference = 1.39, 95% CI 2-sided [0.91 to 1.88]
Statistical Analysis 20: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 7 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.040, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.37, 95% CI 2-sided [-0.71 to -0.02]
Statistical Analysis 21: Comparison: Placebo vs Ibuprofen Sodium; 8 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.20, 95% CI 2-sided [0.71 to 1.69]
Statistical Analysis 22: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 8 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.015, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.44, 95% CI 2-sided [-0.79 to -0.08]

5. Secondary Outcome: Pain Intensity Difference (PID)
Description: PID was derived by subtracting the pain severity score at a given post-dosing time point (pain severity score range 0 [none] to 3 [severe]) from the baseline score (Baseline pain severity score range 2 [moderate] to 3 [severe]). Total possible score range for PID: -1 (worst) to 3 (best).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Units on a scale
  0.25 hours | 0.0 (0.4) | 0.3 (0.5) | 0.1 (0.5)
  0.5 hours | 0.0 (0.5) | 1.0 (0.7) | 0.6 (0.8)
  1 hour | 0.0 (0.7) | 1.5 (0.9) | 1.3 (0.9)
  1.5 hour | 0.0 (0.8) | 1.7 (0.9) | 1.5 (0.9)
  2 hours | 0.0 (0.9) | 1.8 (0.9) | 1.7 (0.9)
  3 hours | 0.0 (0.9) | 1.6 (0.9) | 1.7 (1.0)
  4 hours | 0.1 (1.0) | 1.5 (0.9) | 1.7 (1.0)
  5 hours | 0.0 (1.0) | 1.4 (1.0) | 1.6 (1.0)
  6 hours | -0.0 (0.9) | 1.2 (1.0) | 1.5 (1.1)
  7 hours | -0.0 (0.9) | 0.9 (1.0) | 1.2 (1.1)
  8 hours | -0.0 (0.8) | 0.8 (1.0) | 1.1 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; 0.25 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.30, 95% CI 2-sided [0.13 to 0.46]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 0.25 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.22, 95% CI 2-sided [0.11 to 0.34]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Sodium; 0.5 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.94, 95% CI 2-sided [0.70 to 1.19]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 0.5 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.38, 95% CI 2-sided [0.20 to 0.55]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen Sodium; 1 hour: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.46, 95% CI 2-sided [1.18 to 1.75]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 1 hour: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.017, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.25, 95% CI 2-sided [0.04 to 0.45]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; 1.5 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.67, 95% CI 2-sided [1.39 to 1.96]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 1.5 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.015, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.25, 95% CI 2-sided [0.05 to 0.46]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen Sodium; 2 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.69, 95% CI 2-sided [1.41 to 1.98]
Statistical Analysis 10: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 2 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.362, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.09, 95% CI 2-sided [-0.11 to 0.30]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen Sodium; 3 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.56, 95% CI 2-sided [1.27 to 1.86]
Statistical Analysis 12: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 3 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.472, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.08, 95% CI 2-sided [-0.29 to 0.14]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; 4 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.39, 95% CI 2-sided [1.07 to 1.70]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 4 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.134, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.17, 95% CI 2-sided [-0.40 to 0.05]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen Sodium; 5 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.31, 95% CI 2-sided [1.00 to 1.63]
Statistical Analysis 16: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 5 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.135, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.17, 95% CI 2-sided [-0.40 to 0.05]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen Sodium; 6 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.17, 95% CI 2-sided [0.84 to 1.50]
Statistical Analysis 18: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 6 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.036, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.25, 95% CI 2-sided [-0.49 to -0.02]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen Sodium; 7 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.93, 95% CI 2-sided [0.61 to 1.26]
Statistical Analysis 20: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 7 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.064, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.22, 95% CI 2-sided [-0.46 to 0.01]
Statistical Analysis 21: Comparison: Placebo vs Ibuprofen Sodium; 8 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.85, 95% CI 2-sided [0.52 to 1.18]
Statistical Analysis 22: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 8 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.074, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.22, 95% CI 2-sided [-0.46 to 0.02]

6. Secondary Outcome: Sum of Pain Relief Rating and Pain Intensity Difference (PRID)
Description: PRID was sum of PID and PRR at each post-dosing time point. The overall possible score range, for PRID was -1 (worst) to 7 (best). PID was derived by subtracting the pain severity score at a given post-dosing time point (pain severity score range 0 [none] to 3 [severe]) from the baseline score (Baseline pain severity score range 2 [moderate] to 3 [severe]). Total possible score range for PID: -1 (worst) to 3 (best). PRR was assessed on 5-point categorical pain relief rating scale (0=No relief to 4=Complete relief).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Units on a scale
  0.25 hours | 0.4 (0.9) | 1.1 (1.2) | 0.6 (1.1)
  0.5 hours | 0.6 (1.2) | 3.0 (1.7) | 2.1 (1.8)
  1 hour | 0.7 (1.6) | 4.4 (1.8) | 3.8 (2.0)
  1.5 hours | 0.7 (1.8) | 4.8 (1.8) | 4.3 (2.0)
  2 hours | 0.8 (2.0) | 4.9 (1.8) | 4.7 (2.0)
  3 hours | 0.7 (2.0) | 4.5 (2.0) | 4.7 (2.1)
  4 hours | 0.9 (2.3) | 4.3 (2.1) | 4.8 (2.2)
  5 hours | 0.8 (2.1) | 4.0 (2.2) | 4.4 (2.2)
  6 hours | 0.6 (2.0) | 3.5 (2.2) | 4.1 (2.4)
  7 hours | 0.5 (1.9) | 2.9 (2.3) | 3.5 (2.5)
  8 hours | 0.5 (1.8) | 2.6 (2.3) | 3.2 (2.5)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.65, 95% CI 2-sided [0.26 to 1.04]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.46, 95% CI 2-sided [0.18 to 0.75]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.41, 95% CI 2-sided [1.82 to 3.01]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.91, 95% CI 2-sided [0.48 to 1.34]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.68, 95% CI 2-sided [3.03 to 4.33]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.008, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.64, 95% CI 2-sided [0.17 to 1.11]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 4.06, 95% CI 2-sided [3.40 to 4.72]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 5, analysis 8]; Test type: Superiority or Other; p = 0.017, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.58, 95% CI 2-sided [0.10 to 1.06]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 9]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 4.09, 95% CI 2-sided [3.42 to 4.75]
Statistical Analysis 10: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 5, analysis 10]; Test type: Superiority or Other; p = 0.359, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.22, 95% CI 2-sided [-0.26 to 0.70]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.75, 95% CI 2-sided [3.06 to 4.45]
Statistical Analysis 12: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 5, analysis 12]; Test type: Superiority or Other; p = 0.436, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.20, 95% CI 2-sided [-0.70 to 0.30]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.40, 95% CI 2-sided [2.66 to 4.14]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 5, analysis 14]; Test type: Superiority or Other; p = 0.139, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.40, 95% CI 2-sided [-0.93 to 0.13]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.20, 95% CI 2-sided [2.44 to 3.95]
Statistical Analysis 16: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.144, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.41, 95% CI 2-sided [-0.95 to 0.14]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 17]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.80, 95% CI 2-sided [2.01 to 3.58]
Statistical Analysis 18: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 5, analysis 18]; Test type: Superiority or Other; p = 0.043, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.58, 95% CI 2-sided [-1.15 to -0.02]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.33, 95% CI 2-sided [1.53 to 3.12]
Statistical Analysis 20: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 5, analysis 20]; Test type: Superiority or Other; p = 0.044, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.59, 95% CI 2-sided [-1.16 to -0.02]
Statistical Analysis 21: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.05, 95% CI 2-sided [1.25 to 2.85]
Statistical Analysis 22: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 5, analysis 22]; Test type: Superiority or Other; p = 0.027, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.65, 95% CI 2-sided [-1.23 to -0.08]

7. Secondary Outcome: Time-weighted Sum of Pain Intensity Difference (SPID)
Description: SPID: time-weighted sum of PID over 2, 3, 6 and 8 hours. SPID scores range was -2 (worst) to 6 (best) for SPID 0-2, -3 (worst) to 9 (best) for SPID 0-3, -6 (worst) to 18 (best) for SPID 0-6, -8 (worst) to 24 (best) for SPID 0-8. PID: baseline pain severity score minus pain severity score at a given time point (pain severity score range 0=none to 3=severe; baseline score range 2=moderate to 3=severe). Total score range for PID: -1(worst) to 3 (best).
Time Frame: 0-2, 0-3, 0-6, 0-8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Units on a scale
  SPID 0-2 | 0.1 (1.3) | 2.8 (1.4) | 2.4 (1.5)
  SPID 0-3 | 0.1 (2.1) | 4.4 (2.2) | 4.1 (2.3)
  SPID 0-6 | 0.2 (4.8) | 8.5 (4.7) | 8.9 (5.0)
  SPID 0-8 | 0.1 (6.4) | 10.2 (6.3) | 11.1 (6.7)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; SPID 0-2: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.73, 95% CI 2-sided [2.27 to 3.18]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); SPID 0-2: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.007, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.45, 95% CI 2-sided [0.12 to 0.78]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Sodium; SPID 0-3: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 4.29, 95% CI 2-sided [3.60 to 4.98]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); SPID 0-3: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.144, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.37, 95% CI 2-sided [-0.13 to 0.87]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen Sodium; SPID 0-6: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 8.16, 95% CI 2-sided [6.66 to 9.66]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); SPID 0-6: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.679, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.23, 95% CI 2-sided [-1.31 to 0.85]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; SPID 0-8: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 9.94, 95% CI 2-sided [7.92 to 11.96]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); SPID 0-8: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.367, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.67, 95% CI 2-sided [-2.12 to 0.79]

8. Secondary Outcome: Time-weighted Sum of Pain Relief Rating (TOTPAR)
Description: TOTPAR: time-weighted sum of PRR scores over 2, 3, 6 and 8 hours. TOTPAR score range was 0 (worst) to 8 (best) for TOTPAR 0-2, 0 (worst) to 12 (best) for TOTPAR 0-3, 0 (worst) to 24 (best) for TOTPAR 0-6, 0 (worst) to 32 (best) for TOTPAR 0-8. PRR was evaluated at different time points during the study up to 8 hours, and immediately after taking rescue medication (if necessary). PRR was assessed on a 5-point categorical pain relief rating scale wherein 0=No relief to 4=Complete relief.
Time Frame: 0-2, 0-3, 0-6, 0-8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Units on a scale
  TOTPAR 0-2 | 1.3 (1.8) | 5.2 (1.7) | 4.6 (1.9)
  TOTPAR 0-3 | 2.0 (2.9) | 8.1 (2.7) | 7.6 (2.8)
  TOTPAR 0-6 | 4.2 (6.5) | 15.9 (6.1) | 16.1 (6.1)
  TOTPAR 0-8 | 5.2 (8.4) | 19.5 (8.5) | 20.6 (8.5)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; TOTPAR 0-2: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.95, 95% CI 2-sided [3.32 to 4.59]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); TOTPAR 0-2: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.009, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.62, 95% CI 2-sided [0.16 to 1.07]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Sodium; TOTPAR 0-3: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 6.15, 95% CI 2-sided [5.18 to 7.12]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); TOTPAR 0-3: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.166, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.49, 95% CI 2-sided [-0.21 to 1.20]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen Sodium; TOTPAR 0-6: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 11.67, 95% CI 2-sided [9.54 to 13.81]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); TOTPAR 0-6: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.703, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.30, 95% CI 2-sided [-1.84 to 1.24]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; TOTPAR 0-8: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 14.27, 95% CI 2-sided [11.36 to 17.18]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); TOTPAR 0-8: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.303, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -1.10, 95% CI 2-sided [-3.20 to 1.00]

9. Secondary Outcome: Time-weighted Sum of Pain Relief Rating and Pain Intensity Difference (SPRID)
Description: SPRID: time-weighted sum of PRID over 2, 3, 6 and 8 hours. SPRID score range:-2 (worst) to 14(best) for SPRID 0-2, -3(worst) to 21(best) for SPRID 0-3, -6(worst) to 42(best) for SPRID 0-6, -8(worst) to 56(best) for SPRID 0-8. PRID:sum of PID and PRR at each time point. Total score range for PRID: -1=worst to 7=best. PID:baseline pain severity score minus pain severity score at given time(score range 0=none to 3=severe; baseline score range 2=moderate to 3=severe). Total score range for PID: -1(worst) to 3(best), PRR: scored on 5-point pain relief rating scale(0=No relief to 4=Complete relief).
Time Frame: 0-2, 0-3, 0-6, 0-8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Units on a scale
  SPRID 0-2 | 1.3 (2.9) | 8.0 (3.0) | 7.0 (3.3)
  SPRID 0-3 | 2.1 (4.8) | 12.6 (4.7) | 11.8 (4.9)
  SPRID 0-6 | 4.4 (10.8) | 24.3 (10.4) | 25.0 (10.6)
  SPRID 0-8 | 5.4 (14.1) | 29.8 (14.2) | 31.7 (14.6)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; SPRID 0-2: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 6.68, 95% CI 2-sided [5.60 to 7.76]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); SPRID 0-2: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.007, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.06, 95% CI 2-sided [0.29 to 1.84]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Sodium; SPRID 0-3: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 10.43, 95% CI 2-sided [8.79 to 12.08]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); SPRID 0-3: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.152, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.87, 95% CI 2-sided [-0.32 to 2.05]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen Sodium; SPRID 0-6: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 19.83, 95% CI 2-sided [16.23 to 23.43]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); SPRID 0-6: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.690, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.53, 95% CI 2-sided [-3.12 to 2.07]
Statistical Analysis 7: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); SPRID 0-8 Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and corresponding 95% CI were calculated based on LS mean from the ANOVA model; Test type: Superiority or Other; p = 0.323, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -1.77, 95% CI 2-sided [-5.29 to 1.75]

10. Secondary Outcome: Cumulative Percentage of Participants With Meaningful Relief
Description: Percentage of participants with meaningful relief evaluated by stopping the stopwatch labeled 'meaningful relief' at the moment the participant first began to experience meaningful relief. Stopwatch was active up to 8 hours after dosing or until stopped by the participant, or rescue medication was administered.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Percentage of participants
  0.25 hours | 0.0 | 1.1 | 0.6
  0.5 hours | 4.2 | 28.4 | 16.8
  1 hour | 12.5 | 73.7 | 52.6
  1.5 hours | 14.6 | 87.4 | 69.9
  2 hours | 18.8 | 91.6 | 79.8
  3 hours | 20.8 | 94.7 | 86.7
  4 hours | 20.8 | 94.7 | 87.9
  5 hours | 20.8 | 94.7 | 87.9
  6 hours | 20.8 | 94.7 | 87.9
  7 hours | 20.8 | 95.8 | 87.9
  8 hours | 22.9 | 95.8 | 88.4
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; 0.25 hours-Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on Cochran-Mantel-Haenszel (CMH) adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.490, Cochran-Mantel-Haenszel — p-value was calculated using CMH test which was adjusted for baseline PSR and gender terms. Statistical testing was done at 5% significance level (2-sided); Difference in proportion = 1.01, 95% CI 2-sided [-0.97 to 3.00]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 0.25 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.623, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 0.54, 95% CI 2-sided [-1.88 to 2.95]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Sodium; 0.5 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 24.36, 95% CI 2-sided [13.51 to 35.22]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 0.5 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.023, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 11.82, 95% CI 2-sided [1.15 to 22.48]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen Sodium; 1 hour: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 61.35, 95% CI 2-sided [48.99 to 73.70]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 1 hour: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 21.25, 95% CI 2-sided [9.58 to 32.92]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; 1.5 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 72.65, 95% CI 2-sided [61.59 to 83.71]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 1.5 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 17.44, 95% CI 2-sided [7.83 to 27.06]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen Sodium; 2 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 72.63, 95% CI 2-sided [61.14 to 84.11]
Statistical Analysis 10: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 2 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.013, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 11.70, 95% CI 2-sided [3.47 to 19.93]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen Sodium; 3 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 73.58, 95% CI 2-sided [61.83 to 85.33]
Statistical Analysis 12: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 3 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.041, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 8.01, 95% CI 2-sided [1.27 to 14.75]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; 4 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 73.58, 95% CI 2-sided [61.83 to 85.33]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 4 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.073, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 6.79, 95% CI 2-sided [0.23 to 13.36]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen Sodium; 5 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 73.58, 95% CI 2-sided [61.83 to 85.33]
Statistical Analysis 16: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 5 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.073, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 6.79, 95% CI 2-sided [0.23 to 13.36]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen Sodium; 6 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 73.58, 95% CI 2-sided [61.83 to 85.33]
Statistical Analysis 18: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 6 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.073, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 6.79, 95% CI 2-sided [0.23 to 13.36]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen Sodium; 7 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 74.71, 95% CI 2-sided [63.14 to 86.27]
Statistical Analysis 20: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 7 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.035, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 7.84, 95% CI 2-sided [1.57 to 14.10]
Statistical Analysis 21: Comparison: Placebo vs Ibuprofen Sodium; 8 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 72.61, 95% CI 2-sided [61.05 to 84.17]
Statistical Analysis 22: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); 8 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Advil + Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 7.28, 95% CI 2-sided [1.07 to 13.48]

11. Secondary Outcome: Cumulative Percentage of Participants With Confirmed First Perceptible Relief
Description: Percentage of participants with first perceptible relief was evaluated by stopping a stopwatch labeled 'first perceptible relief' at the moment the participant first began to experience any relief. Stopwatch was active up to 8 hours after dosing or until stopped by the participant, or rescue medication was administered. The first perceptible relief was considered confirmed if the participant also stopped the second stopwatch indicating meaningful relief.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Percentage of participants
  0.25 hours | 6.3 | 26.3 | 12.1
  0.5 hours | 14.6 | 84.2 | 60.7
  1 hour | 20.8 | 94.7 | 84.4
  1.5 hours | 22.9 | 95.8 | 87.3
  2 hours | 22.9 | 95.8 | 87.9
  3 hours | 22.9 | 95.8 | 88.4
  4 hours | 22.9 | 95.8 | 88.4
  5 hours | 22.9 | 95.8 | 88.4
  6 hours | 22.9 | 95.8 | 88.4
  7 hours | 22.9 | 95.8 | 88.4
  8 hours | 22.9 | 95.8 | 88.4
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; 0.25 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 20.01, 95% CI 2-sided [8.79 to 31.24]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 14.35, 95% CI 2-sided [4.26 to 24.43]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 69.53, 95% CI 2-sided [57.67 to 81.40]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 23.45, 95% CI 2-sided [13.16 to 33.75]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 5]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 73.72, 95% CI 2-sided [62.77 to 84.67]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 6]; Test type: Superiority or Other; p = 0.014, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 10.14, 95% CI 2-sided [3.21 to 17.08]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 72.61, 95% CI 2-sided [61.05 to 84.17]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 8]; Test type: Superiority or Other; p = 0.028, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 8.35, 95% CI 2-sided [2.02 to 14.68]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 9]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 72.61, 95% CI 2-sided [61.05 to 84.17]
Statistical Analysis 10: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 10]; Test type: Superiority or Other; p = 0.036, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 7.81, 95% CI 2-sided [1.54 to 14.08]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 11]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 72.61, 95% CI 2-sided [61.05 to 84.17]
Statistical Analysis 12: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 12]; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 7.28, 95% CI 2-sided [1.07 to 13.48]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 72.61, 95% CI 2-sided [61.05 to 84.17]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 14]; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 7.28, 95% CI 2-sided [1.07 to 13.48]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 15]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 72.61, 95% CI 2-sided [61.05 to 84.17]
Statistical Analysis 16: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 16]; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 7.28, 95% CI 2-sided [1.07 to 13.48]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 17]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 72.61, 95% CI 2-sided [61.05 to 84.17]
Statistical Analysis 18: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 18]; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 7.28, 95% CI 2-sided [1.07 to 13.48]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 72.61, 95% CI 2-sided [61.05 to 84.17]
Statistical Analysis 20: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 20]; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 7.28, 95% CI 2-sided [1.07 to 13.48]
Statistical Analysis 21: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 21]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 72.61, 95% CI 2-sided [61.05 to 84.17]
Statistical Analysis 22: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 22]; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 7.28, 95% CI 2-sided [1.07 to 13.48]

12. Secondary Outcome: Time to Treatment Failure
Description: Median time of dropping out of the participants from the study due to lack of efficacy or rescue medication, whichever came first.
Time Frame: 0 to 8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Hours | 1.7 [1.6 to 2.1] | NA [NA to NA] — Data was not summarized as median time to treatment failure was >8 hours for ibuprofen sodium group and therefore 95% CI was not estimable. | NA [NA to NA] — Data was not summarized as median time to treatment failure was >8 hours for ibuprofen (Advil + Motrin IB) group and therefore 95% CI was not estimable.
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p < 0.001, Proportional hazards model — p-value was calculated using PH model with treatment, baseline PSR and gender terms. Statistical testing was done at 5% significance level (2-sided); Hazard Ratio (HR) = 0.13, 95% CI 2-sided [0.08 to 0.22]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p = 0.281, Proportional hazards model — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.79 to 2.22]

13. Secondary Outcome: Cumulative Percentage of Participants With Treatment Failure
Description: Percentage of participants who withdrew from the study due to lack of efficacy or received rescue medication.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Percentage of participants
  0.25 hours | 0.0 | 0.0 | 0.0
  0.5 hours | 0.0 | 0.0 | 0.0
  1 hour | 0.0 | 0.0 | 0.0
  1.5 hours | 25.0 | 1.1 | 2.3
  2 hours | 54.2 | 2.1 | 5.8
  3 hours | 70.8 | 4.2 | 8.1
  4 hours | 70.8 | 9.5 | 8.1
  5 hours | 70.8 | 10.5 | 10.4
  6 hours | 72.9 | 13.7 | 12.1
  7 hours | 77.1 | 20.0 | 16.2
  8 hours | 79.2 | 26.3 | 20.2
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -23.93, 95% CI 2-sided [-36.67 to -11.20]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 8]; Test type: Superiority or Other; p = 0.483, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -1.21, 95% CI 2-sided [-4.12 to 1.70]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 9]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -51.93, 95% CI 2-sided [-65.63 to -38.22]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 10]; Test type: Superiority or Other; p = 0.174, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -3.61, 95% CI 2-sided [-7.97 to 0.75]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 11]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -66.58, 95% CI 2-sided [-79.80 to -53.35]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 12]; Test type: Superiority or Other; p = 0.240, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -3.75, 95% CI 2-sided [-9.38 to 1.89]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -61.36, 95% CI 2-sided [-75.21 to -47.50]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 14]; Test type: Superiority or Other; p = 0.668, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 1.52, 95% CI 2-sided [-5.47 to 8.52]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 15]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -60.31, 95% CI 2-sided [-74.28 to -46.34]
Statistical Analysis 10: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 16]; Test type: Superiority or Other; p = 0.980, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 1.10, 95% CI 2-sided [-7.44 to 7.63]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 17]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -59.28, 95% CI 2-sided [-73.05 to -45.50]
Statistical Analysis 12: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 18]; Test type: Superiority or Other; p = 0.711, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 1.56, 95% CI 2-sided [-6.68 to 9.81]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -56.84, 95% CI 2-sided [-70.84 to -42.85]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 20]; Test type: Superiority or Other; p = 0.445, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 3.72, 95% CI 2-sided [-5.94 to 13.38]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 21]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -52.79, 95% CI 2-sided [-66.77 to -38.81]
Statistical Analysis 16: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 22]; Test type: Superiority or Other; p = 0.256, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 6.05, 95% CI 2-sided [-4.75 to 16.84]

14. Secondary Outcome: Cumulative Percentage of Participants With Complete Relief
Description: Complete relief was defined as a PRR of 4. PRR was assessed on a 5-point categorical pain relief rating scale where 0=No relief to 4=Complete relief.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Percentage of participants
  0.25 hours | 0.0 | 0.0 | 0.0
  0.5 hours | 0.0 | 6.3 | 3.5
  1 hour | 0.0 | 27.4 | 20.8
  1.5 hours | 0.0 | 41.1 | 32.4
  2 hours | 0.0 | 48.4 | 43.9
  3 hours | 0.0 | 52.6 | 54.9
  4 hours | 6.3 | 54.7 | 61.8
  5 hours | 6.3 | 54.7 | 63.0
  6 hours | 6.3 | 54.7 | 63.6
  7 hours | 6.3 | 54.7 | 64.2
  8 hours | 6.3 | 54.7 | 64.2
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p = 0.078, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 6.34, 95% CI 2-sided [1.34 to 11.34]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; p = 0.303, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 2.74, 95% CI 2-sided [-3.01 to 8.49]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 5]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 27.24, 95% CI 2-sided [18.14 to 36.34]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 6]; Test type: Superiority or Other; p = 0.217, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 6.66, 95% CI 2-sided [-4.31 to 17.63]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 41.16, 95% CI 2-sided [31.20 to 51.12]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 8]; Test type: Superiority or Other; p = 0.149, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 8.86, 95% CI 2-sided [-3.33 to 21.04]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 9]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 48.61, 95% CI 2-sided [38.49 to 58.73]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 10]; Test type: Superiority or Other; p = 0.477, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 4.55, 95% CI 2-sided [-8.03 to 17.13]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 11]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 52.81, 95% CI 2-sided [42.63 to 62.99]
Statistical Analysis 10: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 12]; Test type: Superiority or Other; p = 0.739, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -2.14, 95% CI 2-sided [-14.77 to 10.50]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 48.53, 95% CI 2-sided [36.29 to 60.77]
Statistical Analysis 12: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 14]; Test type: Superiority or Other; p = 0.280, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -6.80, 95% CI 2-sided [-19.24 to 5.65]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 15]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 48.53, 95% CI 2-sided [36.29 to 60.77]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 16]; Test type: Superiority or Other; p = 0.202, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -8.01, 95% CI 2-sided [-20.44 to 4.41]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 17]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 48.53, 95% CI 2-sided [36.29 to 60.77]
Statistical Analysis 16: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 18]; Test type: Superiority or Other; p = 0.170, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -8.61, 95% CI 2-sided [-21.02 to 3.80]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 48.53, 95% CI 2-sided [36.29 to 60.77]
Statistical Analysis 18: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 20]; Test type: Superiority or Other; p = 0.140, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -9.23, 95% CI 2-sided [-21.62 to 3.16]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 21]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 48.53, 95% CI 2-sided [36.29 to 60.77]
Statistical Analysis 20: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); [analysis description as in outcome 10, analysis 22]; Test type: Superiority or Other; p = 0.140, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -9.23, 95% CI 2-sided [-21.62 to 3.16]

15. Secondary Outcome: Participant Global Evaluation of Study Medication
Description: Participant global evaluation of study medication was performed at the 8-hour time point or immediately before taking the rescue medication. It was scored on a 6-point categorical scale where 0 = Very poor, 1 = Poor, 2 = Fair, 3 = Good, 4 = Very Good, and 5 = Excellent.
Time Frame: 8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil + Motrin IB)
Number analyzed (Participants) | 48 | 95 | 173
Units on a scale | 1.1 (1.3) | 3.8 (1.0) | 3.7 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; Treatment difference (Ibuprofen sodium - placebo) and the associated CI were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value was calculated using CMH test with modified ridit scores, controlling for baseline PSR and gender terms. Statistical testing was done at 5% significance level (2-sided); Mean Difference (Final Values) = 0.90, 95% CI 2-sided [0.83 to 0.98]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Ibuprofen (Advil + Motrin IB); HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p = 0.667, Proportional hazards model — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.04, 95% CI 2-sided [-0.15 to 0.24]

ADVERSE EVENTS:
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Advil) | Ibuprofen (Motrin IB)
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/95 | 0/86 | 0/87
Other Adverse Events (participants affected / at risk) | 8/48 | 10/95 | 12/86 | 10/87
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | Ibuprofen Sodium (N=95) | Ibuprofen (Advil) (N=86) | Ibuprofen (Motrin IB) (N=87)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Chest discomfort (Cardiac disorders) | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Dyspnoea (Cardiac disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 7 | 6 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2 | 3 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea not otherwise specified (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 2 | 1 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 1 | 0
Hot flush (General disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (General disorders) | 0 | 0 | 0 | 1
Lethargy (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 4 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.